CLINICAL TRIAL: NCT06981494
Title: Dexmedetomidine Versus Dexmedetomidine and Ketamine (Ketodex) Regarding Hemodynamics Stability, Recovery and Postoperative Pain in Ear and Nose Surgeries, A Prospective Randomized Study
Brief Title: Dexmedetomidine Versus Dexmedetomidine and Ketamine (Ketodex) in Ear and Nose Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Madonna Samir Sobhy, Anesthesia resident, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-4-02MS
Record Dates: First submitted 2024-12-26; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Ear and Nose Surgeries With Hypotensive Anaesthesia e.g FESS , MLS , TURBINECTOMY
MeSH Terms: conditions — Microphthalmia, syndromic 7 | interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine Group (D) (Active Comparator): Dexmedetomidine Group (D) :
  We give intravenous the loading and maintenance dose of the general anaesthesia drug Dexmedetomidine
  Loading Dose:
  Dexmedetomidine is usually administered as a loading dose of 0.5 mcg/kg slowly.
  Maintenance Dose:
  After the loading dose, the maintenance infusion rate is typically 0.2 to 0.7 mcg/kg/hour in syringe pump . The exact rate can be adjusted based on the hemodynamics of the patient (blood pressure and heart rate) and the patient's response.
  Interventions: Drug: Dexmedetomidine
- Ketodex Group (Combination of Ketamine and Dexmedetomidine) (K): (Active Comparator): Ketamine Component:
  We give intravenous the loading and maintenance dose of the general anaesthesia drug Dexmedetomidine and ketamine
  Loading Dose:
  Ketamine is typically given at a dose of 0.5 mg/kg as a bolus injection.
  Maintenance Dose:
  A maintenance infusion of 0.2 to 0.5 mg/kg/hour is common to maintain anesthesia in syringe pump.
  Dexmedetomidine Component:
  Loading Dose:
  As with the dexmedetomidine group, a loading dose of 0.5 mcg/kg slowly is administered.
  Maintenance Dose:
  The maintenance infusion rate for dexmedetomidine remains 0.2 to 0.7 µg/kg/hour in syringe pump.
  Interventions: Drug: Dexmedetomidine and ketamine ( Ketodex )

INTERVENTIONS:
Drug: Dexmedetomidine — Loading Dose:
  Dexmedetomidine is usually administered as a loading dose of 0.25 mcg/kg slowly.
  Maintenance Dose:
  After the loading dose, the maintenance infusion rate is typically 0.2 to 0.7 mcg/kg/hour in syringe pump . The exact rate can be adjusted based on the hemodynamics of the patient (blood pressure and heart rate) and the patient's response.
  Arms: Dexmedetomidine Group (D)
Drug: Dexmedetomidine and ketamine ( Ketodex ) — Ketodex Group (Combination of Ketamine and Dexmedetomidine) (K):
  Ketamine Component:
  Loading Dose:
  Ketamine is typically given at a dose of 0.5 mg/kg as a bolus injection.
  Maintenance Dose:
  A maintenance infusion of 0.2 to 0.5 mg/kg/hour is common to maintain anesthesia in syringe pump.
  Dexmedetomidine Component:
  Loading Dose:
  As with the dexmedetomidine group, a loading dose of 0.25 mcg/kg slowly is administered.
  Maintenance Dose:
  The maintenance infusion rate for dexmedetomidine remains 0.2 to 0.7 µg/kg/hour in syringe pump.
  Arms: Ketodex Group (Combination of Ketamine and Dexmedetomidine) (K):

SUMMARY:
The study aims to compare the efficacy, safety and overall effectiveness of dexmedetomidine and dexmedtomidine and ketamine (ketodex) in achieving controlled hypotension during Ear and nose surgeries.

- Assessment the analgesic and sedative role of both drugs.

DETAILED DESCRIPTION:
Comparison regarding the efficacy, safety and overall effectiveness of dexmedetomidine and dexmedtomidine and ketamine (ketodex) in achieving controlled hypotension during Ear and nose surgeries.

* comparison between both drugs in recovery and hemodynamics stability
* Assessment the analgesic and sedative role of both drugs

ELIGIBILITY:
Inclusion Criteria

* Age Range: Patients aged 18-60 years who are scheduled for elective Ear and nose surgeries requiring controlled hypotensive anesthesia.
* ASA Classification: Patients classified as American Society of Anesthesiologists (ASA) physical status I or II.
* Surgical Procedures: Individuals undergoing specific ear and nose surgeries where controlled hypotensive anesthesia is typically indicated.
* Stable Cardiovascular Health: Patients with stable cardiovascular function, without significant history of uncontrolled hypertension , hypotension or ischaemic heart diseases.

Exclusion Criteria

* Severe Cardiovascular Conditions: Patients with severe cardiovascular diseases such as congestive heart failure, uncontrolled hypertension , arrhythmias or ischaemic heart diseases .
* Any cardiac patients.
* Respiratory Conditions: Individuals with significant respiratory conditions like chronic obstructive pulmonary disease (COPD) or severe asthma.
* Drug Allergies: Patients with known hypersensitivity or allergic reactions to dexmedetomidine, ketamine or any other components of the study drugs.
* Pregnancy or Lactation: Pregnant or breastfeeding women, due to potential risks to the fetus or infant.
* Chronic Medication Use: Patients on chronic medications that could interfere with blood pressure regulation or interact with the study drugs (e.g., beta-blockers, MAO inhibitors).
* Patients with chronic liver or renal diseases.
* Psychiatric or Neurological Disorders: Individuals with severe psychiatric or neurological disorders that could impact the study outcomes or the patient's ability to consent.
* Substance Abuse: Patients with a history of substance abuse, particularly involving sedatives or opioids, which could affect anesthesia requirements or recovery.
* Coagulation Disorders: Individuals with coagulation disorders or on anticoagulant therapy, due to the increased risk of bleeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of hemodynmaic stability | 6 months
  Assess Hemodynamic Stability: Compare the hemodynamic stability provided by dexmedetomidine and ketodex, focusing on parameters such as blood pressure and heart rate will be monitored every 5 minutes and we will record the average every 20 minutes intraoperative . This monitoring will help assess the stability of each patient and the safety profile of the anesthetic agents used in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Sohag, Egypt